CLINICAL TRIAL: NCT02483195
Title: The Use of 5mg Finasteride Versus 200mg Spironolactone and Topical 5% Minoxidil in Treating Postmenopausal Female Androgenetic Alopecia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI indicating she was withdrawing her study submission due to lack of funding as of 6/20/2016
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201500433
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Female Androgenetic Alopecia
Keywords: Hair loss; Post Menopausal
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Spironolactone; Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Group (Active Comparator): This group will use a mixed combination of 5% Minoxidil and 200mg Spironolactone for 12 months to be used once daily.
  Interventions: Drug: 5% Minoxidil; Drug: 200mg Spironolactone
- Single Group (Active Comparator): This group will use a mixed combination of 5mg Finasteride with placebo topical preparation for 12 months to be used once daily.
  Interventions: Drug: 5mg Finasteride; Other: Placebo

INTERVENTIONS:
Drug: 5% Minoxidil — This will be a mixed combination of 5% Minoxidil and 200mg Spironolactone to be used once daily.
  Other Names: Rogaine®; Theroxidil®; Minoxidil Topical
  Arms: Combination Group
Drug: 200mg Spironolactone — This will be a mixed combination of 5% Minoxidil and 200mg Spironolactone to be used once daily.
  Other Names: Aldactone®
  Arms: Combination Group
Drug: 5mg Finasteride — This will be a mixed combination of 5mg Finasteride with placebo topical preparation to be used once daily.
  Other Names: Propecia®; Proscar®
  Arms: Single Group
Other: Placebo — This will be a mixed combination of 5mg Finasteride with placebo topical preparation to be used once daily.
  Other Names: placebo topical preparation
  Arms: Single Group

SUMMARY:
The investigators propose to conduct a head-to-head, randomized clinical trial to compare the effectiveness of Minoxidil with Spironolactone and Finasteride in treating postmenopausal females with Androgenetic Alopecia (AGA).

DETAILED DESCRIPTION:
Participants diagnosed with AGA will be randomized into one of the two treatment arms outlined below, and will take the assigned treatment for a total duration of 12 months. Medications will be dispensed by a nurse who is blinded to the participants within each treatment group. Global photograph assessment and participant questionnaires at 0, 4, 8 and 12 months will be the primary means to determine improvement in hair loss.

Compare the following interventions in treating postmenopausal female AGA:

A) Combination 5% Minoxidil and 200mg Spironolactone (Combination Group) B) 5mg Finasteride with placebo topical preparation (Single Group)

ELIGIBILITY:
Inclusion Criteria:

* female
* postmenopausal (>60 years old or with total hysterectomy)
* diagnosed with androgenetic alopecia
* no chemical processing or changes in hair products throughout the study

Exclusion Criteria:

* men
* premenopausal women (<60 or without hysterectomy)
* participants allergic to any of the study medications (minoxidil, finasteride, spironolactone)
* participants with other co-existing forms of alopecia (traction, alopecia areata, or scarring alopecias)
* participants with obstructive uropathy or advanced liver disease
* prior hair loss treatment within the last 6 months
* hair loss from the chemotherapy or other medication-induced alopecia
* Hair loss for greater than 5 years, as medical therapy is unlikely to have much effect at restoring hair follicles inactive for that long of a period.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The Savin Scale will be used to determine hair growth and/or hair loss between the groups. | Change at 0, 4, 8, and 12 months
  This will be based on a photographic scale from D1 to D8. With D1 being minimal disease and D8 being severe alopecia.
The Ludwig Scale will be used to determine hair growth and/or hair loss between the groups. | Change at 0, 4, 8, and 12 months
  This scale is based on the hair loss pattern. Ludwig Scale: Left = pattern 1, middle = pattern 2, right = pattern 3
Alopecia improvement assessment will be used to determine hair growth and/or hair loss between the groups. | Change at 0, 4, 8, and 12 months
  The value will be one of 7 numbers, ranging from -3 to +3. The values will stand for the following:
  * 3: markedly worsened alopecia
  * 2: moderately worsened alopecia
  * 1: slightly worsened alopecia 0: no change in alopecia
    * 1: slightly improved alopecia
    * 2: moderately improved alopecia
    * 3: markedly improved alopecia

CONTACTS AND LOCATIONS:
Overall Officials: Christina L. Mitchell, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States